CLINICAL TRIAL: NCT04239391
Title: Hemoglobin Maintenance in Pediatric ESRD Patients by Ferric Pyrophosphate Citrate (FPC)
Brief Title: Hemoglobin Maintenance in Pediatric ESRD (End-stage Renal Disease) Patients by Ferric Pyrophosphate Citrate (FPC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-22
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-02

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; pediatric; chronic kidney disease; anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — ferric pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triferic via IV and Hemodialysate (Experimental): Upon completion of the Baseline observational periods, all enrolled patients will transition to the interventional period where they will then receive Triferic. The Triferic will be administered via the liquid bicarbonate concentrate at a dialysate concentration of 2 uM or via IV at a dose of 0.1 mg Fe/kg, if the patient does not receive dialysis using liquid bicarbonate, for up to an additional 36 weeks (depending on duration of observational Baseline period). Hgb and CHr will continue to be measured bi-weekly and iron profiles will be obtained at 4 week intervals. In the Triferic phase of the study,changes in ESA dose will be allowed according to the study site existing protocol. IV iron will only be administered if ferritin meets the criteria for iron deficiency. Patients will remain in the interventional period for either 36 or 28 weeks (depending on randomization assignment), at which time a final study visit will take place
  Interventions: Drug: Triferic
- Historic Control Observational Arm (No Intervention): Up to 75 patients will be enrolled in the Observational Arm. Patients who participate in the historical control observational arm will not receive any study medication, but will have Hgb, CHr and serum iron profiles collected at 4 week intervals for up to a total of 44 weeks.

INTERVENTIONS:
Drug: Triferic — Ferric Pyrophosphate Citrate
  Other Names: FPC
  Arms: Triferic via IV and Hemodialysate

SUMMARY:
The main purpose is to determine the safety of Triferic iron administered via dialysate and intravenously in pediatric patients with chronic kidney disease on chronic hemodialysis (CKD-5HD). It is a global, multi- center, open-label study.

DETAILED DESCRIPTION:
This is a global, multi- center, multi dose, open-label study assessing the safety of Triferic iron administered via dialysate and intravenously to pediatric patients (< 18 years of age) receiving chronic hemodialysis (CKD-5HD).

Total participation in the study is approximately 44 weeks and is comprised of a screening visit, baseline, open label treatment, and a follow-up visit.

Upon completion of the respective Baseline observational periods, all patients will transition to the interventional period where they will receive Triferic. The Triferic will be administered via the liquid bicarbonate or via IV. Once patients enter the interventional period, IV iron will only be administered if ferritin <100 µg/L and Hgb decreases by ≥0.5g/dL from the last value obtained in the observational Baseline period. Patients will remain in the interventional period for either 36 or 28 weeks (depending on randomization assignment), at which time a final study visit will take place.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in the study only if all of the following criteria are met:

1. Parents/legal guardians of the patient have the ability to understand the requirements of the study and have demonstrated a willingness to have their child comply with all study procedures by signing an institutional review board-approved informed consent form. Where applicable, assent of the patient has also been obtained for all study procedures prior to any study-related activities.
2. Patient is between 6 months and <18 years of age at screening.
3. Patient has chronic kidney disease receiving in-center hemodialysis at least twice weekly for at least 3 months prior to screening.
4. Patient is receiving adequate hemodialysis as assessed by the investigator and based on a single pool Kt/V measurement >1.2.
5. Patient has a vascular access (tunneled catheter, AV fistula or AV graft) suitable to support blood flows for hemodialysis treatment.
6. Patient has a body mass of ≥11 lbs (5 kg).
7. Patient is iron-replete as measured by a TSAT ≥ 20% and a ferritin >100 µg/L at screening.
8. Patient has a whole blood Hgb concentration of ≥ 9.5 g/dL at screening.
9. If the patient is female, she must be pre-pubertal, have had documented surgical sterilization prior to Baseline admission, or be practicing adequate birth control. All female patients who have reached menarche must have a negative serum pregnancy test during screening. It is the investigator's responsibility to determine whether the patient has adequate birth control for study participation.
10. Patients who have experienced a previous adverse event with IV iron products are eligible to participate in this study if the agent that caused the event is not administered during the Baseline period.

Exclusion Criteria:

A patient will not be eligible for inclusion in the study if any of the following criteria apply:

1. Patient is positive for human immunodeficiency virus (HIV) or hepatitis B by history.
2. Patient is receiving intravenous or oral antibiotics or antifungals for any infectious process. (Prophylactic antibiotics administered on a regular basis are allowed. Patients may enter the study once the infection has cleared.)
3. Patient has evidence of an ongoing active inflammatory process (e.g., systemic lupus erythematosus, acute or chronic active hepatitis, etc.) requiring treatment.
4. Patient has been dosed in an investigational drug study within the 30 days prior to Baseline.
5. Administration of iron containing phosphate binder ferric citrate (Auryxia) or sucroferric oxyhydroxide (Velphoro) within 2 weeks prior to Baseline. (Patient is only eligible if iron based binders are stopped at least 2 weeks prior to Baseline).

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of adverse events of Triferic administration via dialysate and IV in pediatric CKD-5HD patients | 44 weeks
  Incidence and severity of adverse events compared to Baseline.

SECONDARY OUTCOMES:
Assess the ability of Triferic to maintain hemoglobin in pediatric CKD-5HD patients | 44 weeks
  Change from Baseline in hemoglobin concentration
Assess the proportion of patients maintaining hemoglobin between 10.5-12.0 g/dL compared to baseline | 44 weeks
  Proportion of patients maintaining hemoglobin between 10.5 - 12.0 g/dL compared toBaseline
Assess the change in reticulocyte hemoglobin content (CHr). | 44 weeks
  Change from Baseline in reticulocyte hemoglobin content (CHr).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD FACP, Study Director — Rockwell Medical, Inc
Locations (9):
- United States (8):
  - Loma Linda University Hospital, Loma Linda, California
  - Childrens Hospital National Medical Center, Washington D.C., District of Columbia
  - Riley Hospital for Children at Indiana University, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Carolina's Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Health Science Center At San Antonio, San Antonio, Texas
  - Childrens Hospital and Medical Center- Seattle, Seattle, Washington
- University of Puerto Rico School of Medicine, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No